CLINICAL TRIAL: NCT00118846
Title: Phytoestrogens and Progression of Atherosclerosis
Brief Title: Women's Isoflavone Soy Health (WISH) Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH); Office of Research on Women's Health (ORWH) (NIH); Solae, LLC (Industry)
Responsible Party: Principal Investigator, Howard N. Hodis, M.D., Harry J. Bauer and Dorothy Bauer Rawlins Professor of Cardiology, Professor of Medicine, Population and Public Health Sciences, and Molecular Pharmacology and Toxicology, Director, Atherosclerosis Research Unit, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U01AT001653 (NIH); U01AT001653 (NIH); U01AT001653-02S2 (NIH); U01AT001653-02S4 (NIH); U01AT001653-02S5 (NIH)
Record Dates: First submitted 2005-07-07; First posted 2005-07-12 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; Cardiovascular Diseases; Carotid artery intima-media thickness (CIMT); Cognition; Complementary and alternative medicine; Daidzein; Genistein; Glycitein; Intervention; Isoflavones; Menopause; Prevention; Postmenopausal; Randomized controlled study; Soy; Soy Protein; Subclinical Vascular Disease; Ultrasonography; Women
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isoflavone Soy Protein (ISP) Supplementation (Active Comparator): 25 gm soy protein supplementation administered twice daily in equivalent dosages (12.5 gm)
  Interventions: Dietary Supplement: 25 gm soy protein supplement
- Placebo (Placebo Comparator): Milk protein matching placebo administered twice daily in equivalent dosages
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 25 gm soy protein supplement — 25 gm soy protein supplementation administered in equally divided dosage twice daily (12.5 gm)
  Arms: Isoflavone Soy Protein (ISP) Supplementation
Other: Placebo — Milk protein administered twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether soy supplementation can reduce hardening of the arteries and cognitive decline in postmenopausal women.

DETAILED DESCRIPTION:
Heart disease is the leading cause of death among women in the United States. Atherosclerosis, a primary cause of heart disease, accounts for more than 485,000 heart attacks and 370,000 strokes each year in American women. Data indicate that a woman's risk of suffering from an atherosclerosis-related cardiovascular event significantly increases after menopause; this risk may be due to reduced estrogen production associated with menopause. Soy isoflavones are plant compounds that are structurally similar to human estrogen. Evidence suggests that soy supplements may provide the same protection against heart disease as estrogen in postmenopausal women. This study will determine the effects of soy supplementation on subclinical atherosclerosis progression and cognitive decline in postmenopausal women.

In this double-blinded, placebo-controlled trial, a total of 350 postmenopausal women were randomly assigned to receive either soy protein supplementation or placebo twice daily for 2.7 years. The initial 2.5-year treatment period was increased to 3 years. The active product, given as two divided doses, was 25 g soy protein containing 85 mg aglycone weight naturally-occurring isoflavones (150 mg total isoflavone) of genistein 45 mg aglycone weight (80 mg total weight), daidzein 35 mg aglycone weight (60 mg total weight), and glycitein 5 mg aglycone weight (10 mg total weight). The primary trial end point was the rate of change in the right distal common carotid artery intima-media thickness (CIMT) by ultrasonography. Participants underwent ultrasonography at baseline and every six months along with laboratory determinations and clinical measurements. Cognitive assessments were completed at baseline and the final follow-up visit (2.5 years).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined as no vaginal bleeding for at least 1 year and serum estradiol level lower than 20 pg/ml

Exclusion Criteria:

* Signs, symptoms or personal history of cardiovascular disease
* Diabetes mellitus or fasting serum glucose of 126 mg/dL or greater
* Fasting plasma triglyceride of 500 mg/dL or greater
* Serum creatinine greater than 2.0 mg/dL
* Uncontrolled hypertension
* Untreated thyroid disease
* Life expectancy less than 5 years
* Current use of hormone replacement therapy (HRT)
* Soy, nut, or related food allergies
* More than 5 alcohol drinks per day or substance abuse

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2004-04-12 (Actual); Primary Completion 2009-03-19 (Actual); Study Completion 2009-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, M.D., Principal Investigator — Atherosclerosis Research Unit, University of Southern California
Locations (1):
- Atherosclerosis Research Unit, University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Result] Hodis HN, Mack WJ, Kono N, Azen SP, Shoupe D, Hwang-Levine J, Petitti D, Whitfield-Maxwell L, Yan M, Franke AA, Selzer RH; Women's Isoflavone Soy Health Research Group. Isoflavone soy protein supplementation and atherosclerosis progression in healthy postmenopausal women: a randomized controlled trial. Stroke. 2011 Nov;42(11):3168-75. doi: 10.1161/STROKEAHA.111.620831. Epub 2011 Sep 8. PMID 21903957
- [Result] Henderson VW, St John JA, Hodis HN, Kono N, McCleary CA, Franke AA, Mack WJ; WISH Research Group. Long-term soy isoflavone supplementation and cognition in women: a randomized, controlled trial. Neurology. 2012 Jun 5;78(23):1841-8. doi: 10.1212/WNL.0b013e318258f822. PMID 22665144
- [Derived] Lin F, Pa J, Karim R, Hodis HN, Han SD, Henderson VW, St John JA, Mack WJ. Subclinical carotid artery atherosclerosis and cognitive function in older adults. Alzheimers Res Ther. 2022 May 7;14(1):63. doi: 10.1186/s13195-022-00997-7. PMID 35526057
- [Derived] Quaas AM, Kono N, Mack WJ, Hodis HN, Felix JC, Paulson RJ, Shoupe D. Effect of isoflavone soy protein supplementation on endometrial thickness, hyperplasia, and endometrial cancer risk in postmenopausal women: a randomized controlled trial. Menopause. 2013 Aug;20(8):840-4. doi: 10.1097/GME.0b013e3182804353. PMID 23422867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general population through media campaigns.
Pre-assignment Details: 1063 individuals were assessed for eligibility. 713 were not enrolled (660 did not meet inclusion criteria; 53 were eligible but declined to participate). 350 individuals were randomized.
Period: Overall Study
Arm/Group | Isoflavone Soy Protein (ISP) Supplementation | Placebo
Started | 175 | 175
Completed | 162 | 163
Not Completed | 13 | 12
Not completed — Gastrointestinal (GI) intolerance | 3 | 3
Not completed — Started menopausal hormone replacement therapy (HRT) | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Medical condition | 2 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Personal reason | 4 | 5

BASELINE CHARACTERISTICS:
Population: Analysis from participants who had at least one follow-up carotid artery intima-media thickness measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Isoflavone Soy Protein (ISP) Supplementation | Placebo | Total
Number analyzed (Participants) | 162 | 163 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (7.2) | 60.9 (6.9) | 60.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 163 | 325
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (non-Hispanic | 97 | 110 | 207
  Black (non-Hispanic | 12 | 10 | 22
  Hispanic | 31 | 21 | 52
  Asian | 21 | 22 | 43
  Unknown | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 162 | 163 | 325

OUTCOME MEASURES:

1. Primary Outcome: Progression of Subclinical Atherosclerosis
Description: Rate of change in right distal common carotid artery (CCA) far wall intima-media thickness (um per year) in computer image processed B-mode ultrasonograms.
Time Frame: Baseline x 2 and then every 6 months, up to 2.5 years
Population: Rate of change in distal common carotid artery (CCA) far wall intima-media thickness (um per year) in computer image processed B-mode ultrasonograms.
Measure: Mean (95% Confidence Interval); unit: um/year
Arm/Group | Isoflavone Soy Protein (ISP) Supplementation | Placebo
Number analyzed (Participants) | 162 | 163
um/year | 4.77 [3.39 to 6.16] | 5.68 [4.30 to 7.06]
Statistical Analysis 1: Comparison: Isoflavone Soy Protein (ISP) Supplementation vs Placebo; Test type: Superiority; p = 0.35, Mixed Models Analysis; Slope = -0.91, 95% CI 2-sided [-2.86 to 1.05] — Slope = Mean difference in annualized rate of change

2. Secondary Outcome: Change in Neurocognitive Function (Global Cognition)
Description: The specified primary cognitive endpoint compared between treatment groups was change from baseline on a global cognitive composite score calculated as an average of standardized scores for 14 neuropsychological tests weighted by the inverse intertest correlation matrix. Neuropsychological test scores at baseline and follow-up assessments were standardized ([raw score-mean score]/standard deviation) using the baseline means and standard deviations from the entire WISH sample. Each of 3 cognitive composite scores was calculated at baseline and follow-up as the weighted average of the individual donor standardized test scores weighted by the inverse correlation among tests. Change from baseline (endpoint minus baseline cognitive outcome) was computed for each cognitive score (verbal memory, global cognition, executive function). Since the outcome is not a single test but a weighted average of multiple tests, the range is not standardized and there are no established clinical thresholds.
Time Frame: Baseline and 2.5 years
Population: Sample size represents the number of participants with analyzable data collected at baseline and 2.5 years.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Isoflavone Soy Protein (ISP) Supplementation | Placebo
Number analyzed (Participants) | 154 | 159
units on a scale | 0.42 (0.09) | 0.31 (0.08)
Statistical Analysis 1: Comparison: Isoflavone Soy Protein (ISP) Supplementation vs Placebo; Test type: Other; p = 0.36, ANCOVA; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.13 to 0.35]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 2.5 years for each participant.
Description: At each clinic visit, participants were queried about the occurrence of events since their last clinic visit.
Arm/Group | Isoflavone Soy Protein (ISP) Supplementation | Placebo
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/163
Serious Adverse Events (participants affected / at risk) | 69/162 | 65/163
Other Adverse Events (participants affected / at risk) | 162/162 | 163/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isoflavone Soy Protein (ISP) Supplementation (N=162) | Placebo (N=163)
Fibroids Tumor/Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Vaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hysterectomy/Partial/Total/Vaginal (Surgical and medical procedures) | 0 (0) | 1 (1)
Shingles (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Skin tags removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Near/Syncopal/Episode (Nervous system disorders) | 1 (1) | 0 (0)
Colon Cancer/Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
In Situ/Ductal Carcinoma-Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lobular Carcinoma-Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness/Light Headed (Nervous system disorders) | 1 (1) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Cardiac Angiogram (Investigations) | 1 (1) | 0 (0)
Pulmonary Angiogram (Investigations) | 1 (1) | 0 (0)
Eye Infection (Eye disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Seasonal Allergic Reaction/Hay Fever (Immune system disorders) | 1 (1) | 0 (0)
Foreign Object Stuck on throat (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peanut Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Food Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Automobile Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Animal/Insect Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns/Scald (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Soy Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Cold/Flu (Infections and infestations) | 2 (2) | 1 (1)
Sinus Condition/Sinusitis/Sinus Headache/Head Congestion (General disorders) | 1 (1) | 0 (0)
Sore/Irritation/Strep Throat (Infections and infestations) | 1 (1) | 0 (0)
Lower Extremity/Swelling/Stiffness/Pain/Strain/Injury/Cramps/Itching (General disorders) | 1 (1) | 1 (1)
Allergy Problems/Attack (Immune system disorders) | 1 (1) | 0 (0)
Gallbladder Problems/Pain/Attack/Stones (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back Pain/Spasm/Strain/Sprain/Twisted/Hurt/Discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Loss Of Consciousness/Collapsed/Faint/Blacked Out (Nervous system disorders) | 1 (1) | 1 (1)
Muscle Pain/Strain/Sprain/Sore/Spasms/Pulled/Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rectal Bleeding/Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthritis/Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthma Attack/Status Asthmatic/Reoccurrence (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diverticulitis/Diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia/Walking Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hearing Aids/Decrease Hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Headache/Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Knee Tearing/Strain/Tenderness/Swelling/Injury/Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (General disorders) | 1 (1) | 1 (1)
Abdominal Pain/Cramping/Pressure (General disorders) | 1 (1) | 1 (1)
Vomiting/Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea/Loose Stool (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth/Infection/Abscess/Root Canal/Implant/Extraction/Loss/Pain/Dental Work (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip Replacement/Pain/Modification/Revision/Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee Replacement/Surgery (Surgical and medical procedures) | 1 (1) | 2 (2)
Constipation (General disorders) | 1 (1) | 1 (1)
Sciatica/Pain (Nervous system disorders) | 1 (1) | 0 (0)
Hernia Repair/Correction (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary Bladder Problems/Infection/Pressure/Suspension/Spasms/Cramping (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia/Low Hemoglobin/Low Hematocrit/White Blood Cells (Hgb/Hct/WBC) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Jaw Pain/Swelling/ Bone Graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Gums/Implant/Sore/Infection/Surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Body Pain/Swelling/Stiffness (General disorders) | 1 (1) | 0 (0)
Finger Infection/Torn Swollen/Trigger/Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary Problems/Incontinence/Proteinuria/Irritated (Renal and urinary disorders) | 1 (1) | 0 (0)
Cerebral Contusion/Head Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot Problems/Plantar Fasciitis/Foot Drop/Infection/Bones Spur Removal/Bunionectomy/Hammertoe (Surgical and medical procedures) | 2 (2) | 2 (2)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Stomach Burning/Pain/Problems/Tension/Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD Reflux/GI Series/Acid Reflex (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric Ulcers/Bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
H. Pylori (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Bloating/Distension/Gas (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thyroid Gland Swollen/Nodules (Endocrine disorders) | 0 (0) | 1 (1)
Rib Cage Pain/Dislocated (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Bacteria Infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Low Iron Level (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Carpal Tunnel Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Gallbladder Surgery/Laparoscopic Cholecystectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Colon/Colorectal Surgery/Resection/Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Back Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Rectocele Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal Injection/Spinal Epidural (Surgical and medical procedures) | 0 (0) | 1 (1)
Wrist Surgery/Abscess Drained (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal Stenosis Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Cystocele or Vesicocele Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Thigh Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Orthoscopic Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Upper Extremity/Swelling/Stiffness/Pain/Strain/Injury/Cramps/Itching (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isoflavone Soy Protein (ISP) Supplementation (N=162) | Placebo (N=163)
Breast Pain (Reproductive system and breast disorders) | 9 (11) | 3 (3)
Vaginal Spotting/Bleeding/Discharge (Reproductive system and breast disorders) | 12 (18) | 4 (5)
Cataract Surgery/Removal (Eye disorders) | 8 (12) | 5 (6)
Fracture (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (11)
Fall (General disorders) | 8 (8) | 11 (11)
Cold/Flu (Infections and infestations) | 47 (57) | 23 (29)
Sinus Condition/Sinusitis/Sinus Headache/Head Congestion (General disorders) | 12 (17) | 10 (11)
Non-Cardiac Chest Pain (General disorders) | 13 (15) | 13 (19)
Sore/Irritation/Strep Throat (Infections and infestations) | 10 (12) | 3 (3)
Arthritis/Pain (Musculoskeletal and connective tissue disorders) | 13 (16) | 9 (9)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 8 (8)
Urinary Tract Infection (Renal and urinary disorders) | 19 (21) | 5 (5)
Headache/Migraine (Nervous system disorders) | 8 (8) | 6 (6)
Vomiting/Nausea (Gastrointestinal disorders) | 11 (12) | 6 (8)
Lower Extremity/Swelling/Stiffness/Pain/Strain/Injury/Cramps/Itching (General disorders) | 15 (16) | 13 (19)
Upper Extremity/Swelling/Stiffness/Pain/Strain/Injury/Cramps/Itching (General disorders) | 16 (16) | 10 (10)
Diarrhea/Loose Stool (Gastrointestinal disorders) | 2 (3) | 9 (10)
Constipation (Gastrointestinal disorders) | 6 (6) | 15 (17)
Abdominal Bloating/Distension/Gas (Gastrointestinal disorders) | 12 (13) | 16 (20)
Back Pain/Spasm/Strain/Sprain/Twisted/Hurt/Discomfort (Musculoskeletal and connective tissue disorders) | 10 (12) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes